CLINICAL TRIAL: NCT00548951
Title: The Connection Between Sensory Deprivation and Social Withdrawal in Clients of a Long Term Care Facility Living With Alzheimer's Disease and the Effects of a Snoezelen Program.
Brief Title: Alzheimer Patients and the Snoezelen Program
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Queen's University (Other)
Responsible Party: Principal Investigator, Dr. Roumen Milev, Principal Investigator, Queen's University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PSIY-205-05
Record Dates: First submitted 2005-09-12; First posted 2007-10-24 (Estimated); Last update posted 2015-12-16 (Estimated); Status verified 2015-12

CONDITIONS: Dementia
Keywords: Dementia
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): Subject receives Snoezelen sessions once per week.
  Interventions: Other: Snoezelen Room
- 2 (Active Comparator): Subject receives Snoezelen sessions three times per week.
  Interventions: Other: Snoezelen Room
- 3 (Other): Subject receives no sessions per week.
  Interventions: Other: Control

INTERVENTIONS:
Other: Snoezelen Room — Session in a Snoezelen room once per week for 12 weeks
  Arms: 1
Other: Snoezelen Room — Session in a Snoezelen room three times per week for 12 weeks
  Arms: 2
Other: Control — Receive no sessions in a Snoezelen Room.
  Arms: 3

SUMMARY:
To determine the connection between Social Withdrawal and Sensory Deprivation in elderly clients with Alzheimer's Type Dementia (i.e. how providing sensory stimulation might reduce social withdrawal).

DETAILED DESCRIPTION:
The Snoezelen concept or program was originally thought up in Holland and comes from two Dutch words meaning to "sniff and doze". It was first introduced in the Netherlands in the 1970's. The first room was introduced in Snoezelen examines how a group of people react to an area that is private, relaxed and one that they trust. This program will bring out one's sense of taste, touch, smell, sight and hearing just by being in a specially designed room. Trust and relaxation will be looked at by those people with developmental disabilities (those that learn at a slower rate). Snoezelen originated with the belief that everyone needs nerve pulses (senses).

Inside a Snoezelen room you will find, dimmed lights, a relaxed atmosphere and pleasant surroundings, soothing sounds, intriguing aromas, tasty puddings, candies, interesting light effects (fiber optic light spray), comfortable seating, opportunities for interaction and engagement, sense of control over environment, tactile objects (awareness box), bubble tube, solar projector wheel, water fountain, massage pillow, massage tube, tranquility and solitude. The Snoezelen room is an environment in which the primary senses (see, hear, taste, touch) are stimulated all to create an environment that is both relaxing and stimulating. The benefits of Snoezelen change per person but may include some of the following:

* Increased resident and caregiver communication
* Increased awareness and understanding of the environment

The Snoezelen idea: client-controlled, safe comfortable atmosphere and freedom from pressure.

Sensory Deprivation (loss) The average person touches 300 different surfaces every 30 minutes. The average person with a profound disability will likely touch 1-5 surfaces in the same time frame.

ELIGIBILITY:
Inclusion Criteria:

* Residents living at Rideaucrest Home (Long Term Care Facility in Kingston, Ontario);
* Residents having a Mini Mental State Exam with a score of 15 to 27 reflecting mild to moderate dementia;
* Male or female over 65 years of age;
* Resident who are able to leave the terrace;
* Resident who are not actively participating in Life Enrichment Programs;
* Able to provide informed written and signed consent by resident or substitute decision maker.

Exclusion Criteria:

* Suffering from severe life threatening illness with a reasonable expectation of death within the next six month;
* Severe mental disorder in the opinion of the investigator (i.e. bipolar, schizophrenia);
* No recent change in medication(s) during the past four weeks prior to the project;
* Other non-Alzheimer-Type Dementia;
* Residents who suffer from Epilepsy.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 18 (Actual)
Dates: Start 2005-09; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
To evaluate improvement of the residents who are given Snoezelen sessions. | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Roumen V. Milev, MD, Principal Investigator — Queen's University
Locations (1):
- Rideaucrest Home, Kingston, Ontario, Canada